CLINICAL TRIAL: NCT04959721
Title: The Effectiveness of Intra-articular Corticosteroid Injection in Patients With Whiplash-related Neck Pain
Brief Title: Treatment for Whiplash Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Min Cheol Chang (Other)
Responsible Party: Sponsor-Investigator, Min Cheol Chang, Associate Professor, Yeungnam University College of Medicine
Organization: Yeungnam University College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YUMC 2021-06-021
Record Dates: First submitted 2021-06-21; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Cervical Facet Joint Pain
Keywords: Whiplash injury; Cervical facet joint; Chronic pain; Neck pain; Corticosteroid injection
MeSH Terms: conditions — Whiplash Injuries; Chronic Pain; Neck Pain | interventions — Injections; Triamcinolone Acetonide; Bupivacaine; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection group (Experimental): Patients in the injection group will be injected 10 mg (0.25 mL) of triamcinolone acetonide, mixed with 0.25 mL of 0.125% bupivacaine and 0.5 mL of normal saline.
  Interventions: Combination Product: Injection with triamcinolone acetonide, bupivacaine, and normal saline

INTERVENTIONS:
Combination Product: Injection with triamcinolone acetonide, bupivacaine, and normal saline — Triamcinolone acetonide is a synthetic corticosteroid medication used intra-articularly to treat various joint conditions. Bupivacaine is a medication used to decrease feeling in a specific area. In nerve blocks, it is injected around a nerve that supplies the area, or into the spinal canal's epidural space. Saline is most commonly used as a sterile 9 g of salt per litre (0.9%) solution, known as normal saline.
  The procedure will be performed with the patient in a prone position under a C-arm fluoroscopy scanner, with the thorax rests on 2 pillows, flexing the neck maximally, and the head turns 60-90° away from the side of injection. The C-arm tube will be angled cephalad, until it was at a tangent to the cervical facet joint space. A 26-gauge, 90 mm spinal needle will be inserted parallel to the C-arm beam. To confirm intra-articular placement of the needle tip, an arthrogram of the cervical facet joint will be performed by injecting 0.3 mL of contrast.

SUMMARY:
Objective: Cervical facet joint (CFJ) pain is commonly seen after whiplash injuries, and is frequently refractory to physical therapy and oral medication. The investigators will evaluate the effectiveness of intra-articular corticosteroid injection for managing whiplash-related CFJ pain.

Methods: The investigators will recruit 32 patients with chronic and persistent CFJ pain (≥ 3 on the Numeric Rating Scale [NRS]) despite physical therapy and oral medication. Under fluoroscopy guidance, The investigators will inject 10 mg (0.25 mL) of triamcinolone acetonide, mixed with 0.25 mL of 0.125% bupivacaine and 0.5 mL of normal saline. At 1 and 2 months after the injection, pain intensity will be reassessed using the NRS.

ELIGIBILITY:
Inclusion Criteria:

* history of a traffic accident
* ≥ 3-month history of axial cervical pain after the accident without radicular symptoms
* whiplash-associated disorder (WAD) severity of Grade II (neck complaint, decreased range of motion of neck, and point tenderness) at first hospital visit
* failure to respond to physical therapy and oral medication (axial cervical pain of ≥ 3 on the numeric rating scale (NRS 0-10; 0, no pain; 10, worst pain imaginable)
* ≥ 80% temporary pain relief following a diagnostic block with an intra-articular (IA) injection of 0.3 mL of 2% lidocaine

Exclusion Criteria:

* presence of cervical spine fracture, coagulopathy, iodinated contrast allergy, rheumatic disorders, and any uncontrolled medical or psychiatric condition

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Pain before intervention to be assessed with Numeric Rating Scale | The NRS score will be assessed the day before starting the intervention (pre-treatment).
  The investigators will be assessed pain intensity using the NRS score as the primary outcome. Average pain intensity during the 24 hours before NRS assessment will be investigated. The Numeric Rating Scale (NRS) is the simplest and most commonly used numeric scale in which people rate the pain from 0 (no pain) to 10 (worst pain).
Pain after intervention to be assessed with Numeric Rating Scale | The NRS score will be assessed 1 month after the intervention
  The investigators will be assessed pain intensity using the NRS score as the primary outcome. Average pain intensity during the 24 hours before NRS assessment will be investigated. The Numeric Rating Scale (NRS) is the simplest and most commonly used numeric scale in which people rate the pain from 0 (no pain) to 10 (worst pain).
Pain after intervention to be assessed with Numeric Rating Scale | The NRS score will be assessed 2 month after the intervention
  The investigators will be assessed pain intensity using the NRS score as the primary outcome. Average pain intensity during the 24 hours before NRS assessment will be investigated. The Numeric Rating Scale (NRS) is the simplest and most commonly used numeric scale in which people rate the pain from 0 (no pain) to 10 (worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Min Cheol Chang, Study Director — Yuengnam University
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No
Participants' personal information will be stored for 3 years and then destroyed in accordance with relevant regulations. Personal information of individuals is kept strictly confidential and cannot be used for other research without personal consent.

REFERENCES:
- [Background] Crouch R, Whitewick R, Clancy M, Wright P, Thomas P. Whiplash associated disorder: incidence and natural history over the first month for patients presenting to a UK emergency department. Emerg Med J. 2006 Feb;23(2):114-8. doi: 10.1136/emj.2004.022145. PMID 16439739
- [Background] Dory MA. Arthrography of the cervical facet joints. Radiology. 1983 Aug;148(2):379-82. doi: 10.1148/radiology.148.2.6867328.
- [Background] Dussault RG, Nicolet VM. Cervical facet joint arthrography. J Can Assoc Radiol. 1985 Mar;36(1):79-80. PMID 3980558
- [Background] Hove B, Gyldensted C. Cervical analgesic facet joint arthrography. Neuroradiology. 1990;32(6):456-9. doi: 10.1007/BF02426454. PMID 2287370
- [Background] Lim JW, Cho YW, Lee DG, Chang MC. Comparison of Intraarticular Pulsed Radiofrequency and Intraarticular Corticosteroid Injection for Management of Cervical Facet Joint Pain. Pain Physician. 2017 Sep;20(6):E961-E967. PMID 28934800
- [Background] Roy DF, Fleury J, Fontaine SB, Dussault RG. Clinical evaluation of cervical facet joint infiltration. Can Assoc Radiol J. 1988 Jun;39(2):118-20. PMID 2967833